CLINICAL TRIAL: NCT00468611
Title: A Double-Blind, Placebo Controlled Multi-Center Study to Evaluate the Efficacy and Safety of MBP8298 in Subjects With Secondary Progressive Multiple Sclerosis
Brief Title: Efficacy and Safety of MBP8298 in Subjects With Secondary Progressive Multiple Sclerosis
Acronym: MAESTRO-03
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Negative efficacy results of the MAESTRO-01 study
Sponsor: BioMS Technology Corp. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MBP8298-SP-03
Record Dates: First submitted 2007-05-01; First posted 2007-05-03 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Multiple Sclerosis, Secondary Progressive
Keywords: Secondary Progressive Multiple Sclerosis; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — MBP-8298

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: MBP8298
- 2 (Placebo Comparator)
  Interventions: Drug: MBP8298

INTERVENTIONS:
Drug: MBP8298 — 500mg MBP8298 IV every six months for a period of two years

SUMMARY:
This study will assess the efficacy and safety of MBP8298 compared to placebo in subjects with Secondary Progressive Multiple Sclerosis (SPMS)

ELIGIBILITY:
Inclusion Criteria:

* Male of female subjects, 18-65 years of age with a diagnosis of SPMS
* HLA DR2 and/or DR4 positive
* Absence of a relapse in the 3 months prior to baseline
* EDSS of 3.0 - 6.5

Exclusion Criteria:

* Therapy with Beta-interferon, glatiramer acetate within 3 months or mitoxantrone, cyclophosphamide, methotrexate, azathioprine or any immune modulating or immunosuppressive drugs within 6 months of baseline
* Treatment with Tysabri within 2 years of baseline
* Females who are breast feeding, pregnant (pregnancy test at baseline) or not using a medically approved method of contraception regularly

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Time to progression of disease in subjects with SPMS as measured by the EDSS after 24 months of treatment | 24 Months

SECONDARY OUTCOMES:
To assess the safety of MBP8298, degree of change in the EDSS scores, effect of MBP8298 on MRI parameters, difference in relapse rates, effect on MSFC, subject's quality of life (MSQoL54) and fatigue (MFIS) after 24 months of treatment | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Clyde E Markowitz, MD, Principal Investigator — University of Pennsylvania